CLINICAL TRIAL: NCT01770028
Title: Ripple Effect of Lifestyle Intervention During Pregnancy on Partners' Weight
Status: Completed | Type: Observational
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Collaborators: Brown University (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Todd Hagobian, Associate Professor, California Polytechnic State University-San Luis Obispo
Other Study IDs: 1R01HL118208 (NIH)
Record Dates: First submitted 2013-01-08; First posted 2013-01-17 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Obesity
Keywords: Obesity; Pregnancy; Spouse; Weight loss; Behavioral
MeSH Terms: conditions — Obesity; Weight Loss; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 19 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Intervention partners: Partners of pregnant women randomized to lifestyle intervention. Note: There is no intervention in partners of pregnant women.
- Standard care partners: Partners of pregnant women randomized to Standard Care. Note: There is no intervention in partners of pregnant women.

SUMMARY:
The primary aim of the proposed study is to determine whether lifestyle interventions to prevent excessive gestational weight gain in overweight/obese pregnant women have positive "ripple" effects on untreated partners in the home. We hypothesize that partners of pregnant women randomized to the lifestyle intervention, relative to those of standard care, will have greater weight losses through 12-months. Secondary aims examine partner improvements in weight control behaviors, the home environment, and psychosocial parameters.

DETAILED DESCRIPTION:
Lifestyle interventions targeting overweight individuals can produce positive "ripple" effects on untreated overweight partners in the home. Interestingly, ripple effects on partners' weight appear most pronounced when the interventions target women. Women, and mothers in particular, remain the primary "nutritional gatekeepers" of the home. Despite widespread recognition that motherhood is a powerful motivator for behavior changes, no study to date has examined the "ripple" effects of prenatal lifestyle interventions that target mothers' gestational weight gain. The primary aim of the proposed study is to determine whether lifestyle interventions to prevent excessive gestational weight gain in overweight/obese pregnant women have positive "ripple" effects on untreated partners in the home. The proposed study is ancillary to two randomized phase III clinical trials in the LIFE-moms consortium (1U01HL114377-01, PI Phelan; 3U01DK094463-03S1, PIs Pi-Sunyer and Gallagher) that are examining the efficacy of multi-component lifestyle interventions to prevent excessive gestational weight gain in a total of 650 overweight/obese women. In this ancillary study, partners' weight, home environment, and psychosocial behaviors will be assessed when their pregnant partners are ~13 weeks gestation (study entry), 35 weeks gestation and at 6 and 12 months postpartum. We hypothesize that partners of pregnant women randomized to the lifestyle intervention, relative to those of standard care, will have greater weight losses through 12-months. Secondary aims examine partner improvements in weight control behaviors, the home environment, and psychosocial parameters. This project is highly innovative, as it capitalizes on existing funded research and is the first study to examine ripple effects of multicomponent prenatal interventions. The project also has high impact, as pregnancy is a powerful motivator for behavior and environmental changes in the home; and, if positive ripple effects occur, the field of obesity treatment and prevention could move beyond focus on individual level to the often unrecognized interpersonal effects of lifestyle interventions. PUBLIC HEALTH RELEVANCE: This research project will examine whether interventions to prevent excessive gestational weight gain have positive "ripple" effects on the health of untreated partners in the home.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman who self-identifies as sharing an intimate relationship and cohabitating in the home with the pregnant women (enrolled in the parent grant) for the previous 3 months or recently been married and living in the home
* ≥18 years
* willing to provide informed consent/assent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study uses a randomized repeated measures design. Partners will be categorized based on randomized status of their pregnant partner (in the parent grants; NIH 1U01HL114377-01, PI Phelan; NIH 3U01DK094418-01S1, PIs Redman and Martin). Partner participation in the ancillary study will not be mandatory for participation in the parent grant. NOTE: There is no intervention in partners.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2013-01; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in weight of partners of pregnant women | 13 weeks gestation, 35 weeks gestation, 6 months and 12 months postpartum
  Change in weight of partners of pregnant women randomized to the lifestyle intervention, relative to partners of pregnant women of standard care, from 13 weeks gestation to 35 weeks gestation and 6 and 12-months postpartum.

SECONDARY OUTCOMES:
Percent of partners with weight change loss >5%, 10%, and 15% | 13 weeks gestation, 35 weeks gestation, 6 months and 12 months postpartum
Change in calorie and fat intake | 13 weeks gestation, 35 weeks gestation, 6 months and 12 months postpartum
Change in physical activity levels | 13 weeks gestation, 35 weeks gestation, 6 months and 12 months postpartum
Change in sleep patterns and sleep hours | 13 weeks gestation, 35 weeks gestation, 6 months and 12 months postpartum
Change in self-monitoring | 13 weeks gestation, 35 weeks gestation, 6 months and 12 months postpartum
Change in food, exercise and sedentary cues in the home environment | 13 weeks gestation, 35 weeks gestation, 6 months and 12 months postpartum
Change in mood | 13 weeks gestation, 35 weeks gestation, 6 months and 12 months postpartum
Change in dietary restraint | 13 weeks gestation, 35 weeks gestation, 6 months and 12 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Todd A Hagobian, PhD, Principal Investigator — California Polytechnic State University-San Luis Obispo
Locations (3):
- United States (3):
  - California Polytechnic State University, San Luis Obispo, California
  - Columbia University, New York, New York
  - Miriam Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Hagobian TA, Phelan S, Schaffner A, Brannen A, McHugh A, Ashby-Thompson M, Gorin AA, Pi-Sunyer X, Gallagher D, Wing R. Ripple Effect of Lifestyle Interventions During Pregnancy on Untreated Partners' Weight. Obesity (Silver Spring). 2019 May;27(5):733-739. doi: 10.1002/oby.22447. Epub 2019 Apr 8. PMID 30957985